CLINICAL TRIAL: NCT05895955
Title: A Phase I/II Randomized Double Blind Controlled Study to Evaluate the Safety and Immunogenicity of GPO Seasonal Tetravalent Inactivated Split Virion Influenza Vaccine in Healthy Thais
Brief Title: Safety and Immunogenicity of GPO Seasonal Tetravalent Inactivated Split Virion Influenza Vaccine in Healthy Thais
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TetraFluvac TF vaccine
Record Dates: First submitted 2023-05-05; First posted 2023-06-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Influenza
Keywords: Influenza; GPO TetraFluvac Vaccine; TetraFluvac Vaccine; Thais; Thailand; Vaxigrip vaccine; Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Double (Participant, Investigator)
Who Masked: Participant, Investigator
Masking Description: Unblinded study staff, including the site pharmacist, will be responsible for preparing study products (in accordance with the randomly determined assignment), and handling all drug accountability procedures. These personnel will not participate in the other aspects of the clinical trial, to help ensure the integrity of the blind at the site. Unblinded staff will retrieve a participant's randomization assignment after being informed by the PI or designee that a participant is eligible for randomization. They will provide the prefilled 0.5 ml dose of study product based on the participant's randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TetraFluvac TF vaccine (Experimental): 20 participants in phase I study and 200 participants in phase II study will receive a prefilled single dose of 0.5 ml of TetraFluvac TF vaccine will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Interventions: Biological: TetraFluvac TF vaccine
- Vaxigrip vaccine (Active Comparator): 20 participants in phase I study and 50 participants in phase II study will receive a prefilled single dose of 0.5 ml Vaxigrip vaccine (Commercially available seasonal quadrivalent split, manufactured by Sanofi Pasteur, Ltd. France) will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Interventions: Biological: Vaxigrip vaccine

INTERVENTIONS:
Biological: TetraFluvac TF vaccine — The vaccine is a seasonal quadrivalent inactivated split virion influenza vaccine [A/Sydney/5/2021(H1N1) pdm09-like virus and A/Darwin/9/2021 (H3N2)-like virus and B/Austria/1359417/2021 (B/Victoria Lineage)-like virus and B/Phuket/3073/2013 (B/Yamagata lineage)-like virus] produced by The Government Pharmaceutical Organization (GPO), Thailand.
  Each prefilled dose of TetraFluvac TF contains a total of 60 micrograms (μg) hemagglutinin (HA) per 0.5 ml dose (15 μg HA per strain per dose), to be administered by intramuscular (IM) injection.
  Arms: TetraFluvac TF vaccine
Biological: Vaxigrip vaccine — Vaxigrip vaccine is commercially available seasonal quadrivalent inactivated split virion influenza vaccine [A/Sydney/5/2021(H1N1) pdm09-like strain and A/Darwin/9/2021 (H3N2)-like strain and B/Austria/1359417/2021-like strain and B/Phuket/3073/2013-like strain, manufactured by Sanofi Pasteur, Ltd. France.
  Each prefilled dose of Vaxigrip vaccine contains a total of 60 micrograms (μg) hemagglutinin (HA) per 0.5 ml dose (15 μg HA per strain per dose), to be administered by intramuscular (IM) injection.
  Arms: Vaxigrip vaccine

SUMMARY:
The study is aim to evaluate the safety and immunogenicity of one dose TetraFluvac TF vaccine (15 μg HA per strain per dose) of the GPO seasonal quadrivalent inactivated split virion influenza vaccine in healthy adults aged 18 years and above over 90 days post-injection.

DETAILED DESCRIPTION:
This is a double blind randomized study consisting of two phases - Phase I and Phase II.

Phase I of the study A total of 40 healthy participants aged 18 years and above will be enrolled (1:1 ratio, 20 TetraFluvac TF vaccine and 20 Vaxigrip vaccine (Commercially available seasonal quadrivalent split, manufactured by Sanofi Pasteur, Ltd. France)

Phase II of the study A total of 250 healthy participants will be enrolled (4:1 ratio, 200 TetraFluvac TF vaccine and 50 Vaxigrip vaccine (Commercially available seasonal quadrivalent split , manufactured by Sanofi Pasteur, Ltd. France) One dose of the TetraFluvac TF or Commercially available seasonal quadrivalent split vaccine for Southern Hemisphere in 2023 will be given 0.5 ml by intramuscular route.

Total follow-up is 90 days.

The vaccine will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm. After vaccination participants will remain at the clinic for at least 30 minutes to observe for any reactogenicity after immunization.

Blood specimens for immune response will be collected on Day 0 prior to vaccination, Day 28, Day 60, and day 90.

Blood specimen for safety will be collected Day 28 for participants Phase I only for clinical hematology and chemistry.

A DSMB, composed of at least three independent members with expertise in vaccine clinical trials, will be convened to provide additional safety oversight. In Phase I, the DSMB will meet to review all safety profiles of 28 days after immunization. After completing Day 7 of phase I with no safety concern, the screening for phase II can be started. However, the vaccination of phase II will occur after the recommendation of the DSMB.There should be no safety concerns from DSMB meeting for continue Phase II. In Phase II, the DSMB will meet to review all safety profiles after vaccination of 100 participants for completion of Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and above
2. Having Thai ID card or equivalent
3. Able to read and provide written informed consent prior to performance of any study-specific procedure
4. Healthy as defined by no clinically significant acute medical condition, and no chronic medical condition that has not been controlled within 90 days of randomization, as determined by medical history, physical examination, screening laboratory test results, and clinical assessment of the investigator.
5. All hematology, biochemistry and urine analysis are within normal range or of no clinical significance (not higher than 1.5 time of normal value without any clinical finding from history and physical examination)

Exclusion Criteria:

1. Known history of egg allergy
2. Having had recently influenza infection confirmed as H1N1, H3N2, or Flu B within 3 months preceding enrollment to the trial
3. Vaccination against influenza in the past 6 months preceding enrollment to the trial
4. History of bronchial asthma, chronic lung diseases, chronic rhinitis
5. History of immunodeficiency state
6. History of immunosuppression < 6 months prior to immunization
7. History of anaphylactic or other allergic reactions to influenza vaccine or any vaccine component or excipient (e.g. gentamicin or thimerosal)
8. Acute infectious with fever > 38 degree Celsius and noninfectious diseases (within 72 hours) preceding enrollment in the trial
9. The participants who have been taking immunoglobulin products or have had a blood transfusion during past 3 months before the beginning of the experiment
10. Participation in other research study
11. Pregnancy or plan to become pregnant for 60 days after enrollment or breast feeding
12. Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
13. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled, or could interfere with the evaluation of the vaccine
14. Employee of any person employed by the Sponsor, the contract research organization (CRO), the PI, study site personnel, or site.
15. Any test for HIV, HBsAg, Hep C antibody shows positive results with clinically significance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2023-11-04 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of Solicited local adverse events post-vaccination. | 30-minutes after vaccination
  Frequency of solicited reportable local adverse events (pain or tenderness, limitation arm movement, erythema, swelling or induration)
Number and percentage of Solicited local adverse events post-vaccination. | day 1
  Frequency of solicited reportable local adverse events (pain or tenderness, limitation arm movement, erythema, swelling or induration)
Number and percentage of Solicited local adverse events post-vaccination. | day 2
  Frequency of solicited reportable local adverse events (pain or tenderness, limitation arm movement, erythema, swelling or induration)
Number and percentage of Solicited local adverse events post-vaccination. | day 3
  Frequency of solicited reportable local adverse events (pain or tenderness, limitation arm movement, erythema, swelling or induration)
Number and percentage of Solicited local adverse events post-vaccination. | day 4
  Frequency of solicited reportable local adverse events (pain or tenderness, limitation arm movement, erythema, swelling or induration)
Number and percentage of Solicited local adverse events post-vaccination. | day 5
  Frequency of solicited reportable local adverse events (pain or tenderness, limitation arm movement, erythema, swelling or induration)
Number and percentage of Solicited local adverse events post-vaccination. | day 6
  Frequency of solicited reportable local adverse events (pain or tenderness, limitation arm movement, erythema, swelling or induration)
Number and percentage of Solicited local adverse events post-vaccination. | day 7
  Frequency of solicited reportable local adverse events (pain or tenderness, limitation arm movement, erythema, swelling or induration)
Number and percentage of Solicited systemic adverse events post-vaccination. | 30-minutes after vaccination
  Frequency of solicited reportable systemic adverse events (fever, chill, headache, rhinorrhea, fatigue or malaise, myalgia, arthralgia, rash, nausea or vomiting, diarrhea)
Number and percentage of Solicited systemic adverse events post-vaccination. | day 1
  Frequency of solicited reportable systemic adverse events (fever, chill, headache, rhinorrhea, fatigue or malaise, myalgia, arthralgia, rash, nausea or vomiting, diarrhea)
Number and percentage of Solicited systemic adverse events post-vaccination. | day 2
  Frequency of solicited reportable systemic adverse events (fever, chill, headache, rhinorrhea, fatigue or malaise, myalgia, arthralgia, rash, nausea or vomiting, diarrhea)
Number and percentage of Solicited systemic adverse events post-vaccination. | day 3
  Frequency of solicited reportable systemic adverse events (fever, chill, headache, rhinorrhea, fatigue or malaise, myalgia, arthralgia, rash, nausea or vomiting, diarrhea)
Number and percentage of Solicited systemic adverse events post-vaccination. | day 4
  Frequency of solicited reportable systemic adverse events (fever, chill, headache, rhinorrhea, fatigue or malaise, myalgia, arthralgia, rash, nausea or vomiting, diarrhea)
Number and percentage of Solicited systemic adverse events post-vaccination. | day 5
  Frequency of solicited reportable systemic adverse events (fever, chill, headache, rhinorrhea, fatigue or malaise, myalgia, arthralgia, rash, nausea or vomiting, diarrhea)
Number and percentage of Solicited systemic adverse events post-vaccination. | day 6
  Frequency of solicited reportable systemic adverse events (fever, chill, headache, rhinorrhea, fatigue or malaise, myalgia, arthralgia, rash, nausea or vomiting, diarrhea)
Number and percentage of Solicited systemic adverse events post-vaccination. | day 7
  Frequency of solicited reportable systemic adverse events (fever, chill, headache, rhinorrhea, fatigue or malaise, myalgia, arthralgia, rash, nausea or vomiting, diarrhea)
Number and percentage of participants with unsolicited adverse events | day 0 up to day 90
  All unsolicited adverse events during 90 days will be analysed in terms of number and percentage and relationship to study vaccine
  Number and percentage of participants with unsolicited adverse events
Number and percentage of participants with AESI | day 0 up to day 90
  Number and percentage of participants with AESI
Number and percentage of participants with Medically-Attended Adverse Event | day 0 up to day 90
  Number and percentage of participants with Medically-Attended Adverse Event
Number and percentage of participants with Serious Adverse Event | day 0 up to day 90
  Number and percentage of participants with Serious Adverse Event

SECONDARY OUTCOMES:
Antihemagglutinin antibody titer changed from baseline. | day 28
  Seroconversion is defined as a 4-fold rise in HI titer in post-immunization serum relative to pre-immunization serum, or if pre-immunization serum had an undetectable titer (<1:10), attainment of a post-immunization titer of ≥1:40.
Antihemagglutinin antibody titer changed from baseline. | day 60
  Seroconversion is defined as a 4-fold rise in HI titer in post-immunization serum relative to pre-immunization serum, or if pre-immunization serum had an undetectable titer (<1:10), attainment of a post-immunization titer of ≥1:40.
Antihemagglutinin antibody titer changed from baseline. | day 90
  Seroconversion is defined as a 4-fold rise in HI titer in post-immunization serum relative to pre-immunization serum, or if pre-immunization serum had an undetectable titer (<1:10), attainment of a post-immunization titer of ≥1:40.
Geometric mean of immune response changed from baseline | day 28
  The analysis was performed only as intention-to-treat (ITT). The antibody titer values were transformed into log10 titers for calculation of the GMT at every time of assessment
Geometric mean of immune response changed from baseline | day 60
  The analysis was performed only as intention-to-treat (ITT). The antibody titer values were transformed into log10 titers for calculation of the GMT at every time of assessment
Geometric mean of immune response changed from baseline | day 90
  The analysis was performed only as intention-to-treat (ITT). The antibody titer values were transformed into log10 titers for calculation of the GMT at every time of assessment

CONTACTS AND LOCATIONS:
Overall Officials: PUNNEE PITISUTTITHUM, M.D, Principal Investigator — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No